CLINICAL TRIAL: NCT04090658
Title: Phase I, Observer-blind, Safety, Reactogenicity and Immunogenicity Study of GSK's Respiratory Syncytial Virus (RSV) Vaccine GSK3844766A in Japanese Subjects Aged 60-80 Years
Brief Title: A Study to Test GlaxoSmithKline's (GSK) Respiratory Syncytial Virus RSV Candidate Vaccine's Safety and Immune Response in Japanese Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 209699
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Results first posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2021-12

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSV_PreF3_AS01B Group (Experimental): Subjects aged 60 to 80 years received 2 doses of the investigational adjuvanted RSV_PreF3 vaccine (GSK3844766A), at Day 1 and Day 61, by intramuscular (IM) injection into the deltoid region of the non-dominant arm preferably.
  Interventions: Biological: RSV_PreF3 Vaccine (GSK3844766A) adjuvanted with AS01B
- Placebo Group (Placebo Comparator): Subjects aged 60 to 80 years received 2 doses of placebo as control, at Day 1 and Day 61, by IM injection into the deltoid region of the non-dominant arm preferably.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: RSV_PreF3 Vaccine (GSK3844766A) adjuvanted with AS01B — Subjects aged 60 to 80 years received 2 doses of the investigational adjuvanted RSV_PreF3 vaccine (GSK3844766A), at Day 1 and Day 61, by intramuscular (IM) injection into the deltoid region of the non-dominant arm preferably.
  Arms: RSV_PreF3_AS01B Group
Drug: Placebo — Subjects aged 60 to 80 years received 2 doses of placebo as control, at Day 1 and Day 61, by IM injection into the deltoid region of the non-dominant arm preferably.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of 2 doses of GSK Biologicals' RSV candidate vaccine adjuvanted with AS01B for the prevention of lower respiratory tract diseases caused by RSV in ethnic Japanese adults 60-80 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performance of any study specific procedure.
* A male or female between, and including, 60 and 80 years of age at the time of the first vaccination.
* Subjects with residence status allowing free mixing with general community or in an assisted-living facility that provides minimal assistance, such that the subject is primarily responsible for self-care and activities of daily living, may be enrolled.
* Japanese ethnic origin (defined as having been born in Japan with four ethnic Japanese grandparents and able to speak Japanese).
* Subject satisfying screening requirements.

Exclusion Criteria:

Medical conditions

* Any medical condition that in the judgment of the investigator would make IM injection unsafe.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Serious or unstable chronic illness. Patients with chronic stable conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, are allowed to participate in this study.
* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* History of any neurological disorders or seizures.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by the investigator based on medical history, physical examination or laboratory screening tests.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Lymphoproliferative disorder and malignancy within 5 years.
* At screening: Hematology parameters (complete blood cell count [red blood cells, WBC], white blood cells differential count [lymphocytes, neutrophils and eosinophils], platelets count or hemoglobin level) and/or biochemistry parameters (creatinine, blood urea nitrogen or liver enzymes [ALT or AST]) outside the normal laboratory ranges, unless the laboratory abnormalities are considered not clinically significant by the investigator.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine during the period starting 30 days before the first dose of study vaccine (Day -29 to Day 1), or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of study vaccine administration, with the exception of inactivated and subunit influenza vaccines which can be administered up to 14 days before or from 30 days after each study vaccination.
* Previous vaccination with an RSV vaccine.
* Known previous administration of a vaccine containing MPL, QS-21 and/or MF59.
* Planned administration of GSK's Herpes Zoster vaccine marketed as Shingrix or an adjuvanted recombinant varicella zoster virus envelope gE subunit vaccine [HZ/su] within 180 days after the second dose of the study vaccine.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 6 months prior to the first vaccine dose. For corticosteroids, this will mean prednisone (≥ 20 mg/day, or equivalent). Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first dose of study vaccine or planned administration during the study period.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).

Other exclusions

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Body mass index greater than 40 kg/m^2.
* Planned move to a location that will prohibit participating in the trial until study end.
* Bedridden subjects.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Kotb S, Haranaka M, Folschweiller N, Nakanwagi P, Verheust C, De Schrevel N, David MP, Mesaros N, Hulstrom V. Safety and immunogenicity of a respiratory syncytial virus prefusion F protein (RSVPreF3) candidate vaccine in older Japanese adults: A phase I, randomized, observer-blind clinical trial. Respir Investig. 2023 Mar;61(2):261-269. doi: 10.1016/j.resinv.2022.11.003. Epub 2023 Jan 12. PMID 36641341

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (5.0) | 67.2 (4.2) | 66.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Adverse Events (AEs) After First Dose of Vaccination
Description: Assessed solicited local AEs at injection site are pain, erythema and swelling. Any erythema/swelling is scored with a diameter larger than (>) 20 millimeters (mm).
Time Frame: During a 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) after first dose of vaccination administered at Day 1
Population: The analysis was performed on the Exposed Set that included all subjects with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  Erythema | 1 | 0
  Pain | 17 | 1
  Swelling | 2 | 0

2. Primary Outcome: Number of Subjects With Solicited Local AEs After Second Dose of Vaccination
Description: Assessed solicited local AEs at injection site are pain, erythema and swelling. Any erythema/swelling was scored with a diameter larger than (>) 20 millimeters (mm).
Time Frame: During a 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) after second dose of vaccination administered at Day 61
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  Erythema | 0 | 0
  Pain | 17 | 4
  Swelling | 0 | 0

3. Primary Outcome: Number of Subjects With Solicited General AEs After First Dose of Vaccination
Description: Assessed solicited general AEs solicited were: arthralgia; fatigue; fever (any temperature greater than or equal to 38.0 °C - the preferred location for measuring temperature being the oral cavity); gastrointestinal symptoms (including nausea, vomiting, diarrhea and/or abdominal pain); headache; myalgia and shivering.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  Arthralgia | 1 | 0
  Fatigue | 9 | 2
  Fever | 0 | 0
  Gastrointestinal symptoms | 1 | 1
  Headache | 2 | 2
  Myalgia | 6 | 0
  Shivering | 1 | 0

4. Primary Outcome: Number of Subjects With Solicited General AEs After Second Dose of Vaccination
Description: Assessed solicited general AEs solicited are: arthralgia; fatigue; fever (any temperature greater than or equal to 38.0 °C - the preferred location for measuring temperature being the oral cavity); gastrointestinal symptoms including (nausea, vomiting, diarrhea and/or abdominal pain); headache; myalgia and shivering.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  Arthralgia | 5 | 0
  Fatigue | 9 | 1
  Fever | 4 | 0
  Gastrointestinal symptoms | 0 | 1
  Headache | 5 | 1
  Myalgia | 5 | 1
  Shivering | 4 | 0

5. Primary Outcome: Number of Subjects With Unsolicited AEs After Any Vaccination
Description: An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited AE.
Time Frame: During a 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) after any vaccination (across doses)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants | 7 | 6

6. Primary Outcome: Number of Subjects Presenting Change From Baseline in Hematology and Biochemistry With Respect of Normal Laboratory Ranges, After First Vaccine Dose When Compared to Day 1
Description: Assessed hematological laboratory parameters include basophils, eosinophils, erythrocytes, hemoglobin, lymphocytes, monocytes, neutrophils, platelets, white blood cells. Biochemical laboratory parameters include alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine, urea nitrogen and uric acid. Categories reported when comparing Day 1 (pre-vaccination dose 1=baseline) and Day 8 hematological and biochemical laboratory results are defined as follows: <parameter>-<range at baseline>-<range at timing> (e.g. ALT-Within-Within). Ranges level being classified as below, within or above the normal ranges.
Time Frame: At 7 days after the first vaccine dose (i.e. at Day 8 versus Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  ALT-Above-Above: number analyzed (Participants) | 1 | 0
  ALT-Above-Above | 1 | 0
  ALT-Within-Within: number analyzed (Participants) | 19 | 20
  ALT-Within-Within | 19 | 20
  AST-Within-Above | 0 | 1
  AST-Within-Within | 20 | 19
  Basophils-Within-Within | 20 | 20
  Creatinine-Within-Below | 1 | 0
  Creatinine-Within-Within | 19 | 20
  Eosinophils-Below-Below: number analyzed (Participants) | 5 | 2
  Eosinophils-Below-Below | 3 | 1
  Eosinophils-Below-Within: number analyzed (Participants) | 5 | 2
  Eosinophils-Below-Within | 2 | 1
  Eosinophils-Within-Below: number analyzed (Participants) | 15 | 18
  Eosinophils-Within-Below | 2 | 1
  Eosinophils-Within-Within: number analyzed (Participants) | 15 | 18
  Eosinophils-Within-Within | 13 | 17
  Erythrocytes-Below-Below: number analyzed (Participants) | 0 | 1
  Erythrocytes-Below-Below | 0 | 1
  Erythrocytes-Within-Below: number analyzed (Participants) | 20 | 19
  Erythrocytes-Within-Below | 2 | 2
  Erythrocytes-Within-Within: number analyzed (Participants) | 20 | 19
  Erythrocytes-Within-Within | 18 | 17
  Hemoglobin-Below-Below: number analyzed (Participants) | 0 | 1
  Hemoglobin-Below-Below | 0 | 1
  Hemoglobin-Within-Below: number analyzed (Participants) | 20 | 19
  Hemoglobin-Within-Below | 0 | 1
  Hemoglobin-Within-Within: number analyzed (Participants) | 20 | 19
  Hemoglobin-Within-Within | 20 | 18
  Lymphocytes-Within-Within | 20 | 20
  Monocytes-Below-Below: number analyzed (Participants) | 3 | 1
  Monocytes-Below-Below | 2 | 0
  Monocytes-Below-Within: number analyzed (Participants) | 3 | 1
  Monocytes-Below-Within | 1 | 1
  Monocytes-Within-Below: number analyzed (Participants) | 17 | 19
  Monocytes-Within-Below | 1 | 0
  Monocytes-Within-Within: number analyzed (Participants) | 17 | 19
  Monocytes-Within-Within | 16 | 19
  Neutrophils-Below-Below: number analyzed (Participants) | 1 | 0
  Neutrophils-Below-Below | 1 | 0
  Neutrophils-Within-Within: number analyzed (Participants) | 19 | 20
  Neutrophils-Within-Within | 19 | 20
  Platelets-Within-Within | 20 | 20
  Urea Nitrogen-Above-Within: number analyzed (Participants) | 1 | 0
  Urea Nitrogen-Above-Within | 1 | 0
  Urea Nitrogen-Within-Within: number analyzed (Participants) | 19 | 20
  Urea Nitrogen-Within-Within | 19 | 20
  Uric Acid-Above-Above: number analyzed (Participants) | 3 | 0
  Uric Acid-Above-Above | 1 | 0
  Uric Acid-Above-Within: number analyzed (Participants) | 3 | 0
  Uric Acid-Above-Within | 2 | 0
  Uric Acid-Within-Above: number analyzed (Participants) | 17 | 20
  Uric Acid-Within-Above | 1 | 1
  Uric Acid-Within-Below: number analyzed (Participants) | 17 | 20
  Uric Acid-Within-Below | 1 | 0
  Uric Acid-Within-Within: number analyzed (Participants) | 17 | 20
  Uric Acid-Within-Within | 15 | 19
  White Blood Cells-Below-Below: number analyzed (Participants) | 1 | 2
  White Blood Cells-Below-Below | 1 | 0
  White Blood Cells-Below-Within: number analyzed (Participants) | 1 | 2
  White Blood Cells-Below-Within | 0 | 2
  White Blood Cells-Within-Below: number analyzed (Participants) | 19 | 18
  White Blood Cells-Within-Below | 1 | 0
  White Blood Cells-Within-Within: number analyzed (Participants) | 19 | 18
  White Blood Cells-Within-Within | 18 | 18

7. Primary Outcome: Number of Subjects Presenting Change From Baseline in Hematology and Biochemistry With Respect of Normal Laboratory Ranges, After Second Vaccine Dose When Compared to Day 61
Description: Assessed hematological laboratory parameters include basophils, eosinophils, erythrocytes, hemoglobin, lymphocytes, monocytes, neutrophils, platelets, white blood cells. Biochemical laboratory parameters include alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine, urea nitrogen and uric acid. Categories reported when comparing Day 61 (pre-vaccination dose 2=baseline) and Day 68 hematological and biochemical laboratory results are defined as follows: <parameter>-<range at baseline>-<range at timing> (e.g. ALT-Within-Within). Ranges level being classified as below, within or above the normal ranges.
Time Frame: At 7 days after the second vaccine dose (i.e at Day 68 versus Day 61)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  ALT-Within-Within | 20 | 20
  AST-Within-Above | 0 | 1
  AST-Within-Within | 20 | 19
  Basophils-Within-Within | 20 | 20
  Creatinine-Below-Below: number analyzed (Participants) | 0 | 1
  Creatinine-Below-Below | 0 | 1
  Creatinine-Within-Above: number analyzed (Participants) | 20 | 19
  Creatinine-Within-Above | 0 | 1
  Creatinine-Within-Below: number analyzed (Participants) | 20 | 19
  Creatinine-Within-Below | 1 | 0
  Creatinine-Within-Within: number analyzed (Participants) | 20 | 19
  Creatinine-Within-Within | 19 | 18
  Eosinophils-Below-Within: number analyzed (Participants) | 1 | 0
  Eosinophils-Below-Within | 1 | 0
  Eosinophils-Within-Above: number analyzed (Participants) | 19 | 20
  Eosinophils-Within-Above | 1 | 0
  Eosinophils-Within-Within: number analyzed (Participants) | 19 | 20
  Eosinophils-Within-Within | 18 | 20
  Erythrocytes-Below-Below: number analyzed (Participants) | 1 | 3
  Erythrocytes-Below-Below | 0 | 3
  Erythrocytes-Below-Within: number analyzed (Participants) | 1 | 3
  Erythrocytes-Below-Within | 1 | 0
  Erythrocytes-Within-Below: number analyzed (Participants) | 19 | 17
  Erythrocytes-Within-Below | 1 | 1
  Erythrocytes-Within-Within: number analyzed (Participants) | 19 | 17
  Erythrocytes-Within-Within | 18 | 16
  Hemoglobin-Below-Within: number analyzed (Participants) | 1 | 0
  Hemoglobin-Below-Within | 1 | 0
  Hemoglobin-Within-Below: number analyzed (Participants) | 19 | 20
  Hemoglobin-Within-Below | 0 | 2
  Hemoglobin-Within-Within: number analyzed (Participants) | 19 | 20
  Hemoglobin-Within-Within | 19 | 18
  Lymphocytes-Within-Within | 20 | 20
  Monocytes-Below-Below: number analyzed (Participants) | 2 | 0
  Monocytes-Below-Below | 2 | 0
  Monocytes-Within-Below: number analyzed (Participants) | 18 | 20
  Monocytes-Within-Below | 2 | 0
  Monocytes-Within-Within: number analyzed (Participants) | 18 | 20
  Monocytes-Within-Within | 16 | 20
  Neutrophils-Below-Below: number analyzed (Participants) | 1 | 1
  Neutrophils-Below-Below | 1 | 1
  Neutrophils-Within-Below: number analyzed (Participants) | 19 | 19
  Neutrophils-Within-Below | 0 | 1
  Neutrophils-Within-Within: number analyzed (Participants) | 19 | 19
  Neutrophils-Within-Within | 19 | 18
  Platelets-Within-Within | 20 | 20
  Urea Nitrogen-Within-Within | 20 | 20
  Uric Acid-Above-Above: number analyzed (Participants) | 0 | 1
  Uric Acid-Above-Above | 0 | 1
  Uric Acid-Below-Below: number analyzed (Participants) | 1 | 0
  Uric Acid-Below-Below | 1 | 0
  Uric Acid-Within-Above: number analyzed (Participants) | 19 | 19
  Uric Acid-Within-Above | 1 | 1
  Uric Acid-Within-Below: number analyzed (Participants) | 19 | 19
  Uric Acid-Within-Below | 1 | 0
  Uric Acid-Within-Within: number analyzed (Participants) | 19 | 19
  Uric Acid-Within-Within | 17 | 18
  White Blood Cells-Below-Below: number analyzed (Participants) | 3 | 1
  White Blood Cells-Below-Below | 1 | 0
  White Blood Cells-Below-Within: number analyzed (Participants) | 3 | 1
  White Blood Cells-Below-Within | 2 | 1
  White Blood Cells-Within-Below: number analyzed (Participants) | 17 | 19
  White Blood Cells-Within-Below | 0 | 1
  White Blood Cells-Within-Within: number analyzed (Participants) | 17 | 19
  White Blood Cells-Within-Within | 17 | 18

8. Primary Outcome: Number of Subjects With Any Grade 3 Non-serious AEs (Solicited and Unsolicited) After First Dose of Vaccination
Description: A Grade 3 AE is any AE assessed as severe, i.e. which prevents normal, everyday activities. In adults, such an AE would, for example, prevent attendance at work and would necessitate the administration of corrective therapy.
Time Frame: During a 30-day follow-up period (i.e., on the day of vaccination at Day 1, and 29 subsequent days) after first vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  Any adverse event | 0 | 0
  General adverse event | 0 | 0
  Local adverse event | 0 | 0

9. Primary Outcome: Number of Subjects With Any Grade 3 Non-serious AEs (Solicited and Unsolicited) After Second Dose of Vaccination
Description: as for outcome 8
Time Frame: During a 30-day follow-up period (i.e., on the day of vaccination at Day 61, and 29 subsequent days) after second vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  Any adverse event | 2 | 0
  General adverse event | 1 | 0
  Local adverse event | 1 | 0

10. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) up to 30 Days After the Second Vaccination
Description: A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity.
Time Frame: From Day 1 up to 30 days after the second vaccination (Day 91)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants | 0 | 1

11. Primary Outcome: Number of Subjects With Any Potential Immune-mediated Diseases (pIMDs) up to 30 Days After the Second Vaccination
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology
Time Frame: From Day 1 up to 30 days after the second vaccination (Day 91)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

12. Secondary Outcome: Humoral Immune Response With Respect to Components of the Investigational Vaccine in Terms of Neutralizing Antibody Titers Against RSV- Serotype A
Description: Serological assays for the determination of functional antibodies against RSV-A were performed by neutralization assay. Anti RSV-A neutralizing antibody titers are given as geometric mean titers (GMTs) and expressed as Estimated Dose: serum dilution giving a 60% reduction of the signal compared to a control without serum (ED60). The cut-off of the assay is 18 ED60.
Time Frame: At pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), on the day of second vaccination (Day 61) and 30 days post-Dose 2 (Day 91)
Population: The analysis was performed on the Per Protocol Set (PPS) that included all subjects who received at least 1 dose of the study treatment to which they were randomized and had post-vaccination data, minus subjects with protocol deviations that led to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Titers
  Day 1 | 727.3 [445.6 to 1187.3] | 656 [464.7 to 926.2]
  Day 31 | 5315 [3452.8 to 8181.5] | 582.3 [372.1 to 911.2]
  Day 61 | 4382.8 [2828.1 to 6792.1] | 646.1 [442.6 to 943.1]
  Day 91 | 4605.2 [3031.2 to 6996.4] | 529.9 [352.4 to 796.9]

13. Secondary Outcome: Humoral Immune Response With Respect to Components of the Investigational Vaccine in Terms of RSVPreF3-specific Immunoglobulin G (IgG) Antibody Concentrations
Description: The detection and the quantification of total IgG antibodies directed against RSVPreF3 in human serum samples are based on an indirect enzyme-linked immunosorbent assay (ELISA). Anti RSVPreF3 antibody concentration is given in geometric mean concentration (GMC) and is expressed in ELISA Laboratory Units per milliliter (ELU/mL). The assay cut-off is 25 ELU/mL.
Time Frame: as for outcome 12
Population: The analysis was performed on the PPS that included all subjects who received at least 1 dose of the study treatment to which they were randomized and had post-vaccination data, minus subjects with protocol deviations that led to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
ELU/mL
  Day 1 | 6676.7 [4490 to 9928.2] | 7090.2 [5123.8 to 9811.4]
  Day 31 | 85282.4 [66071.9 to 110078.4] | 7242.6 [5534.1 to 9478.6]
  Day 61 | 54076.9 [40417.7 to 72352.2] | 5625.9 [4322.5 to 7322.3]
  Day 91 | 61110.7 [45959 to 81257.6] | 5515.7 [4240.2 to 7174.8]

14. Secondary Outcome: Number of Subjects With Any SAEs, up the End of Follow-up Study Period (Month 14)
Description: as for outcome 10
Time Frame: From Day 1 up to the end of follow-up period (Month 14)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants | 0 | 1

15. Secondary Outcome: Number of Subjects Reporting pIMDs up to the End of Follow-up Study Period (Month 14)
Description: as for outcome 11
Time Frame: From Day 1 up to the end of follow-up period (Month 14)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

16. Secondary Outcome: Number of Subjects With Respiratory Tract Infection (RTI) Episodes Reported During RTI Surveillance
Description: The number of RTI cases is provided by group. Reported categories are "RSV+ RTI" (= RTI episode tested as RSV positive by quantitative reverse transcription polymerase chain reaction (qRT-PCR) on nasal/throat swab collected at assessment visit) and "RSV- RTI" (= RTI episode tested as RSV negative by qRT-PCR on nasal/throat swab collected at assessment visit).
Time Frame: During the RSV seasons from Day 1 to Month 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
Number analyzed (Participants) | 20 | 20
Participants
  RSV + RTI | 0 | 0
  RSV - RTI | 1 | 1

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during the 7-day follow-up period after each vaccination. Unsolicited AEs were collected during the 30-day follow-up period after any vaccination. SAEs were collected during the whole study period, from Day 1 till Month 14.
Arm/Group | RSV_PreF3_AS01B Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 19/20 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV_PreF3_AS01B Group (N=20) | Placebo Group (N=20)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV_PreF3_AS01B Group (N=20) | Placebo Group (N=20)
Injection site pain (General disorders) | 18 (34) | 4 (5)
Fatigue (General disorders) | 13 (18) | 2 (3)
Chills (General disorders) | 6 (6) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 0 (0)
Injection site swelling (General disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 0 (0)
Headache (Nervous system disorders) | 7 (8) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT04090658/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT04090658/SAP_001.pdf